CLINICAL TRIAL: NCT05313711
Title: Study of Use of 'Photographic Rhinometry' Following Derm and Mohs Micrographic Surgery for Skin Cancers: A Follow-up Study
Brief Title: Photographic Rhinometry Following Derm/Mohs Surgery for Skin Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1-075-21
Record Dates: First submitted 2021-11-03; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dermatological surgeons and patients routinely notice alterations in nasal shape and size following surgery and reconstruction. There is no uniform approach to objectively measure these changes. Anthropometric measurements are routinely used in rhinoplasty to assess outcomes, but they are time consuming and have not been reported as being used by dermatological surgeons. Soft-tissue measurements in profile photographs have been demonstrated to be useful for objective measurement of nasal change following surgery. This is a follow up study of the pilot study to assess the feasibility of photographic rhinometry as an objective tool, and (ii) to quantify changes following common dermatological surgical procedures on the nose. This follow-up study will aim to recruit a larger population sample to better quantify some of the changes occurring post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male and female participants
* Type of cancer: Undergoing surgery for removal of Basal Cell Carcinoma (BCC), Squamous Cell Carcinoma (SCC))

Exclusion Criteria:

* Cases unable to consent to participation in the study
* Patients who are unable to complete the study assessments
* Patients below 18 years of age
* Patients undergoing surgery for other types of skin cancer

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 68 participants undergoing surgery for removal of Basal Cell Carcinoma (BCC), Squamous Cell Carcinoma (SCC).
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to quantify changes following common dermatological surgical procedures on the nose. | "baseline, pre-intervention/procedure/surgery" and "immediately after the intervention/procedure/surgery"
  Photographs will be taken with a camera in fixed zoom setting with a ruler placed in different anatomical sites before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Rajpara, MD, Principal Investigator — NHS Grampian
Locations (2):
- United Kingdom (2):
  - Burnside House, Foresterhill Health Campus, Cornhill Road,, Aberdeen
  - The Hillingdon Hospitals NHS Foundation Trust, Uxbridge

IPD SHARING:
Plan to Share IPD: No